CLINICAL TRIAL: NCT06214455
Title: The Effect of a No-added Sugar Diet, Time-restricted Eating and Periodic Water Fasting on Long COVID Symptoms
Brief Title: Diet and Fasting for Long COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Northwest University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-06-PNWU
Record Dates: First submitted 2023-01-03; First posted 2024-01-19 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Long Covid19; Long COVID
Keywords: COVID-19; fasting; diet
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm AB (Diet then Fasting) (Experimental): 2 week baseline with a low sugar diet and 10-12 eating window
  Treatment A: Eat a low sugar diet, 10-12 hour eating window for four weeks
  Treatment B: Eat a low sugar diet, 8 hour eating window, 23 to 60 hour fast once a week for four weeks
  Interventions: Other: Low sugar diet and 10-12 hour eating window; Other: Low sugar diet, 8 hour eating window and fasting
- Arm BA (Fasting then Diet) (Experimental): 2 week baseline with a low sugar diet and 10-12 eating window
  Treatment B: Eat a low sugar diet, 8 hour eating window, 23 to 60 hour fast once a week for four weeks
  Treatment A: Eat a low sugar diet, 10-12 hour eating window for four weeks
  Interventions: Other: Low sugar diet and 10-12 hour eating window; Other: Low sugar diet, 8 hour eating window and fasting

INTERVENTIONS:
Other: Low sugar diet and 10-12 hour eating window — Low sugar diet and 10-12 hour eating window for four weeks
Other: Low sugar diet, 8 hour eating window and fasting — Low sugar diet, 8 hour eating window and a 36-60 hour fast once per week for four weeks.

SUMMARY:
This cross-over study will assess a no added sugar diet, a restricted daily eating window, and one or two full day water fasts to determine if there is an effect on self-reported symptoms of Long Covid (PASC).

DETAILED DESCRIPTION:
This remote study will use a cross-over design to test a diet change plus a 10-12 hour eating window (Treatment A) compared to a diet change, an 8-hour eating window, and one 36 or 60 hour fast per week (Treatment B). Both potential Treatment A and potential Treatment B are 4 weeks in duration. To be eligible, subjects must have a minimum of five common long COVID-19 symptoms. The fasting will limit food intake but not water intake. There will be a two-week run-in with weekly surveys of patient-reported symptoms and severity. The subjects will be randomly assigned to Group AB or to Group BA. Since the water fasts are at the beginning of the week (with symptoms surveyed at the end of the week) there is a 5-6 day washout and then a cross-over to the other treatment for Group BA. A Likert 0-4 scale is used to track the severity of 28 of the most common patient-reported symptoms each week. An additional 30 symptoms are also tracked. Subjects are asked to follow a no-added sugar diet for the entire 10 weeks of the study.

ELIGIBILITY:
Inclusion Criteria

* Adult (18-69 years old)
* Five or more common Long Covid symptoms
* Free from fever > 100F and known bacterial and parasitic infections
* Must indicate willingness to limit certain supplements and report all medications.
* Must indicate willingness to make significant dietary changes - and limit daily eating to an 8 or 10 hour window.
* Must indicate willingness to attempt 36 hr or 60 hr water fasts each week for 4 weeks.
* Have a valid email address and phone number
* Reside in the United States
* Be able to read and to communicate in English
* Must indicate willingness to avoid "extra" supplements such as Fish Yes Oil, Cod liver Oil, Krill Oil, MCT oil, Coconut Oil, Tumeric/Curcumin, Berberine, Quercetin (> 500 mg), Red Yeast Rice, French Marine Bark extract, Red Sage, Ginko biloba, Oregano Oil, Peppermint Oil, Black seed oil, Cinnamon bark extract, Elderberry, Stinging Nettle, Milk Thistle, Monolaurin, Vendicinals 9, Tollovid, QuadraMune and all Probiotics.
* Must indicate willingness to avoid certain nutraceuticals such as Zinc (more than 25 mg), Arginine, Glutamine, Palmitoylethanolamide (PEA), Alpha Lipoic Acid, L Carnitine and Taurine during the study period.
* Must indicate willingness to avoid longevity supplements such as NAD+, Niacin, NMN, Nicotinamide Riboside, Spermidine and Fisetin during the study period.
* Must indicate willingness to halt Olive oil consumption greater than 1 tsp daily during the study period.

Exclusion Criteria:

* Likely COVID-19 or SARS-CoV-2 infection < 45 days before enrollment
* Body Mass Index (BMI) must be 20 or greater
* Past history of an eating disorder.
* Previously fasted more than 18 hours with Long COVID
* Currently doing intermittent fasting
* Pregnant or breast-feeding
* Severe pulmonary disease requiring supplemental oxygen
* Partial loss of vision due to macular degeneration
* Any recent (90 days) history of malignancies, fractures, surgery, radiation, chemo, anesthesia, or traumas
* Diagnosed with Type I or Type II Diabetes
* Previous Autoimmune condition
* Heart condition (Coronary artery disease, Heart valve disease, Heart No failure, Stroke)
* Pre-pandemic Arrythmia
* Liver disease
* Previous Chronic Health Conditions that did not fully resolve (Includes ME/CFS, Lyme Disease, and Fibromyalgia)
* Prescription anticoagulation medication that cannot be halted during the study period. Brilinta (ticagrelor), Plavix (clopidogrel), Coumadin, Warfarin etc.
* High Cholesterol medications that cannot be halted or reduced during the study period (Fenofibrate, Statins > 10 mg)
* Anti-inflammatories or immunosuppressants such as Steroids, Low dose Naltrexone (LDN), Maraviroc, Remicade/Infliximab or Colchicine that cannot be halted during the study period
* Metformin, Ivermectin, or peptides such as BCP-157 that cannot be halted during the study period

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change in Long COVID Symptom Scores during Treatment A vs Treatment B | 4 weeks for each treatment
  Long COVID Symptom Severity Scores are calculated from weekly surveys using a (0-4) severity scale for each of 28 patient-reported symptoms commonly found in Long COVID. The symptom severity values are summed for each participant. That severity subtotal is then added to the number of 30 additional symptoms that were reported.
Change in number of Long COVID symptoms during Treatment A vs Treatment B | 4 weeks for each treatment (delta from week 6 to week 2 or from week 10 to week 6)
  The total number of patient-reported symptoms is calculated from the weekly symptom surveys. The value at the end of the 4 week treatment period is subtracted from the value at the beginning of the 4 week treatment period.

SECONDARY OUTCOMES:
Change in Long COVID Symptom Scores during the 10 week trial | 10 weeks (delta from week 10 to week 0)
  Long COVID Symptom Severity Scores are calculated from weekly surveys using a (0-4) severity scale for each of 28 patient-reported symptoms commonly found in Long COVID. The symptom severity values are summed for each participant. That severity subtotal is then added to the number of 30 additional symptoms that were reported.
Change in number of Long COVID symptoms during the 10 week trial | 10 weeks (delta from week 10 to week 0)
  The total number of patient-reported symptoms is calculated from the weekly symptom surveys. The value at the end of the 4 week treatment period is subtracted from the value at the beginning of the 4 week treatment period.
Number of participants With Serious and Concerning Adverse Events | 2 week baseline, 4 weeks for Treatment A, 4 weeks for Treatment B, 10 weeks of the study
  All adverse events will be medically reviewed and judged to be; not related, possibly related, or definitely related to the treatment intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Novack, PhD, Principal Investigator — Pacific Northwest University of Health Sciences
Locations (2):
- United States (2):
  - Remote trial - anyone residing in the United States, Boulder, Colorado
  - Pacific Northwest University, Yakima, Washington

IPD SHARING:
Plan to Share IPD: No
No current plan to share data with other researchers.

REFERENCES:
- [Background] Stein SR, Ramelli SC, Grazioli A, Chung JY, Singh M, Yinda CK, Winkler CW, Sun J, Dickey JM, Ylaya K, Ko SH, Platt AP, Burbelo PD, Quezado M, Pittaluga S, Purcell M, Munster VJ, Belinky F, Ramos-Benitez MJ, Boritz EA, Lach IA, Herr DL, Rabin J, Saharia KK, Madathil RJ, Tabatabai A, Soherwardi S, McCurdy MT; NIH COVID-19 Autopsy Consortium; Peterson KE, Cohen JI, de Wit E, Vannella KM, Hewitt SM, Kleiner DE, Chertow DS. SARS-CoV-2 infection and persistence in the human body and brain at autopsy. Nature. 2022 Dec;612(7941):758-763. doi: 10.1038/s41586-022-05542-y. Epub 2022 Dec 14. PMID 36517603
- [Background] Cheung CCL, Goh D, Lim X, Tien TZ, Lim JCT, Lee JN, Tan B, Tay ZEA, Wan WY, Chen EX, Nerurkar SN, Loong S, Cheow PC, Chan CY, Koh YX, Tan TT, Kalimuddin S, Tai WMD, Ng JL, Low JG, Yeong J, Lim KH. Residual SARS-CoV-2 viral antigens detected in GI and hepatic tissues from five recovered patients with COVID-19. Gut. 2022 Jan;71(1):226-229. doi: 10.1136/gutjnl-2021-324280. Epub 2021 Jun 2. No abstract available. PMID 34083386
- [Background] Davis HE, Assaf GS, McCorkell L, Wei H, Low RJ, Re'em Y, Redfield S, Austin JP, Akrami A. Characterizing long COVID in an international cohort: 7 months of symptoms and their impact. EClinicalMedicine. 2021 Aug;38:101019. doi: 10.1016/j.eclinm.2021.101019. Epub 2021 Jul 15. PMID 34308300
- [Background] Diebold SS, Kaisho T, Hemmi H, Akira S, Reis e Sousa C. Innate antiviral responses by means of TLR7-mediated recognition of single-stranded RNA. Science. 2004 Mar 5;303(5663):1529-31. doi: 10.1126/science.1093616. Epub 2004 Feb 19. PMID 14976261
- [Background] Girdhar K, Powis A, Raisingani A, Chrudinova M, Huang R, Tran T, Sevgi K, Dogus Dogru Y, Altindis E. Viruses and Metabolism: The Effects of Viral Infections and Viral Insulins on Host Metabolism. Annu Rev Virol. 2021 Sep 29;8(1):373-391. doi: 10.1146/annurev-virology-091919-102416. PMID 34586876
- [Background] Gold JE, Okyay RA, Licht WE, Hurley DJ. Investigation of Long COVID Prevalence and Its Relationship to Epstein-Barr Virus Reactivation. Pathogens. 2021 Jun 17;10(6):763. doi: 10.3390/pathogens10060763. PMID 34204243
- [Background] Hannan MA, Rahman MA, Rahman MS, Sohag AAM, Dash R, Hossain KS, Farjana M, Uddin MJ. Intermittent fasting, a possible priming tool for host defense against SARS-CoV-2 infection: Crosstalk among calorie restriction, autophagy and immune response. Immunol Lett. 2020 Oct;226:38-45. doi: 10.1016/j.imlet.2020.07.001. Epub 2020 Jul 10. PMID 32659267
- [Background] Heil F, Hemmi H, Hochrein H, Ampenberger F, Kirschning C, Akira S, Lipford G, Wagner H, Bauer S. Species-specific recognition of single-stranded RNA via toll-like receptor 7 and 8. Science. 2004 Mar 5;303(5663):1526-9. doi: 10.1126/science.1093620. Epub 2004 Feb 19. PMID 14976262
- [Background] Kim H, Rebholz CM, Hegde S, LaFiura C, Raghavan M, Lloyd JF, Cheng S, Seidelmann SB. Plant-based diets, pescatarian diets and COVID-19 severity: a population-based case-control study in six countries. BMJ Nutr Prev Health. 2021 Jun 7;4(1):257-266. doi: 10.1136/bmjnph-2021-000272. eCollection 2021. PMID 34308134
- [Background] Koepke L, Hirschenberger M, Hayn M, Kirchhoff F, Sparrer KM. Manipulation of autophagy by SARS-CoV-2 proteins. Autophagy. 2021 Sep;17(9):2659-2661. doi: 10.1080/15548627.2021.1953847. Epub 2021 Jul 19. PMID 34281462
- [Derived] Bunker T, Horne BD, Baldwin MD, Sorrells R, Turner S, Laube L, Solomon A, Horne LA, Novack J. Intermittent fasting and a no-sugar diet for Long COVID symptoms: a randomized crossover trial. Sci Rep. 2025 Jul 29;15(1):27563. doi: 10.1038/s41598-025-07461-0. PMID 40730806

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT06214455/Prot_SAP_000.pdf